CLINICAL TRIAL: NCT01795820
Title: Platelet Aggregation During Pharmacological Shift From Clopidogrel to Ticagrelor in Patients With Acute Coronary Syndrome
Brief Title: Platelet Aggregation During the Shift From Clopidogrel to Ticagrelor
Acronym: SHIFT-OVER
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University Magna Graecia (Other)
Responsible Party: Principal Investigator, Ciro Indolfi, Head of Department (Dipartimento di Scienze Mediche e Chirurgiche), University Magna Graecia
Allocation: Randomized | Model: Parallel | Masking: Single
Other Study IDs: SHIFT-OVER
Record Dates: First submitted 2013-02-04; First posted 2013-02-21 (Estimated); Last update posted 2013-02-21 (Estimated); Status verified 2013-02

CONDITIONS: Acute Coronary Syndrome
Keywords: ticagrelor; clopidogrel; platelet aggregation
MeSH Terms: conditions — Acute Coronary Syndrome | interventions — Ticagrelor

STUDY DESIGN:
Who Masked: Participant

ARMS (2):
- Group 1 (no loading) (Other): Patients allocated to this group will not receive a loading dose of ticagrelor. In other words, clopidogrel 75 mg/die will be administered until the day before the pharmacological shift (study start), while ticagrelor 90 mg bis in die will be administered from the day of the pharmacological shift on.
  Interventions: Drug: no loading with Ticagrelor
- Group 2 (loading) (Other): Patients allocated to this group will receive a loading dose of ticagrelor. In other words, clopidogrel 75 mg/die will be administered until the day before the pharmacological shift (study start). On the very day of the pharmacological shift, patients allocated in Group 2 will receive Ticagrelor 180 mg (loading dose) on the morning and Ticagrelor 90 mg on the evening, while ticagrelor 90 mg bis in die will be administered from the day after the pharmacological shift on.
  Interventions: Drug: loading with Ticagrelor

INTERVENTIONS:
Drug: loading with Ticagrelor — Patients allocated in the two study arms will receive the same anti platelet treatment, except for the administration of the loading dose, which will be only administered to patients allocated in Group 2
  Arms: Group 2 (loading)
Drug: no loading with Ticagrelor — Patients allocated in the two study arms will receive the same anti platelet treatment, except for the administration of the loading dose, which will be only administered to patients allocated in Group 2.
  In other words, patients randomized to this group (group 1) will not receive a loading dose of ticagrelor during the passage from clopidogrel to ticagrelor.
  Arms: Group 1 (no loading)

SUMMARY:
Antiplatelet therapy with ticagrelor is currently indicated for treatment of patients presenting with acute coronary syndrome. Such therapy is started with the administration of a loading dose in patients which are not yet under treatment with P2Y12 inhibitors (antiplatelet agents). However it is unknown whether a loading dose is needed to maintain a satisfactory inhibition of platelet aggregation in patients who are already treated with a previous generation P2Y12 inhibitor (clopidogrel) during the passage to the newer compound ticagrelor. For this reason aim of the present study is to evaluate the levels of platelet aggregation during the pharmacological shift from clopidogrel to ticagrelor performed with or without a loading starting dose of the newer drug.

ELIGIBILITY:
Inclusion Criteria:

* Acute Coronary Syndrome
* Current dual anti platelet treatment with ASA and Clopidogrel

Exclusion Criteria:

* No coronary revascularization within the previous six months
* Ongoing therapy with ticagrelor, prasugrel or ticlopidine before enrollment
* No treatment with glycoprotein IIb/IIIa inhibitors within the previous 6 days
* Patients which are known to be no responders to Clopidogrel
* Known neoplastic or autoimmune disease
* Liver cirrhosis
* Severe pulmonary disease
* Known disorder of Haemostasis
* Previous Stroke
* Ongoing pregnancy
* Therapy with any inhibitor of P450 Cytochrome until 15 days before enrollment
* Low platelet count or Hb<10 g/dl

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Actual)
Dates: Start 2012-11; Primary Completion 2013-01 (Actual)

PRIMARY OUTCOMES:
Platelet aggregation | 2 hours
  Platelet aggregation is measured by means of Multiple Electrode Aggregometry (MEA) and Light Transmission Aggregometry (LTA).

SECONDARY OUTCOMES:
30-days clinical events | 30 days
  major adverse cardiac events (MACE) and bleedings will be evaluated per telephone call at 30 days

CONTACTS AND LOCATIONS:
Overall Officials: Ciro Indolfi, MD, Principal Investigator — Magna Graecia University
Locations (1):
- Magna Graecia University, Catanzaro, Calabria, Italy

REFERENCES:
- [Derived] Caiazzo G, De Rosa S, Torella D, Spaccarotella C, Mongiardo A, Giampa S, Micieli M, Palella E, Gulletta E, Indolfi C. Administration of a loading dose has no additive effect on platelet aggregation during the switch from ongoing clopidogrel treatment to ticagrelor in patients with acute coronary syndrome. Circ Cardiovasc Interv. 2014 Feb;7(1):104-12. doi: 10.1161/CIRCINTERVENTIONS.113.000512. Epub 2014 Jan 21. PMID 24449597
- See also: Related Info — http://dsmc.unicz.it/